CLINICAL TRIAL: NCT01894815
Title: Escitalopram and Transcranial Direct Current Stimulation in Major Depressive Disorder: a Double-blind, Placebo-controlled, Randomized, Non-inferiority Trial
Brief Title: Escitalopram, Placebo and tDCS in Depression: a Non-inferiority Trial
Acronym: ELECT-TDCS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Brain & Behavior Research Foundation (Other)
Responsible Party: Principal Investigator, Andre Brunoni, MD, PhD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ELECT-TDCS; FAPESP 2012/20911-5 (Other Grant/Funding Number: FAPESP 2012/20911-5)
Record Dates: First submitted 2013-07-03; First posted 2013-07-10 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-12

CONDITIONS: Major Depressive Disorder; Major Depressive Disorder, Recurrent, Unspecified; Major Depressive Disorder, Single Episode, Unspecified
Keywords: major depressive disorder; major depression; depressive disorder; major depressive episode
MeSH Terms: conditions — Depressive Disorder, Major; Recurrence; Depressive Disorder | interventions — Escitalopram; Transcranial Direct Current Stimulation; Clinical Trials as Topic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Active tDCS / placebo pill (Experimental): transcranial direct current stimulation, using the parameters specified in Interventions.
  Interventions: Device: transcranial direct current stimulation
- Sham tDCS / escitalopram (Active Comparator): Escitalopram oxalate (Reconter), 10mg/day (first 3 weeks) and 20mg/day (week 3 to week 10).
  Interventions: Drug: Escitalopram oxalate
- Sham tDCS / placebo pill (Placebo Comparator): For sham tDCS, the device is automatically turned off after 30 second of stimulation and remains turned off during the 30-min session.
  For placebo pill, the pill has the same size, taste and color than escitalopram, and placebo and escitalopram will be provided in identical bottles, differing only according to a random-generated number placed in the label.
  Interventions: Other: Sham tDCS + Placebo Pill

INTERVENTIONS:
Drug: Escitalopram oxalate — The investigators will use 10mg and 20mg pills. The investigators will up-titrate escitalopram from 10 to 20mg/day according to the patient tolerability. The maximum dose (20mg/day) is sought to be achieved at week 3.
  Other Names: Reconter
  Arms: Sham tDCS / escitalopram
Device: transcranial direct current stimulation — The anode will be applied over the F3 area and the cathode over the F4 area. The current dose is 2mA, current density is 0.8 A/m2. Electrodes will be 5x5cm in size. The investigators will apply 15 daily, consecutive tDCS sessions (excluding weekends) and after that one session per week until the primary endpoint.
  Other Names: tDCS - Soterix Medical Device for Clinical Trials
  Arms: Active tDCS / placebo pill
Other: Sham tDCS + Placebo Pill — This group receives sham tDCS and placebo pill.
  Arms: Sham tDCS / placebo pill

SUMMARY:
Major depressive disorder (MDD) is a common psychiatric condition, mostly treated with antidepressant drugs, which are limited for issues such as refractoriness and adverse effects. In this context, the investigators investigate a non-pharmacological treatment known as transcranial direct current stimulation (tDCS). To prove that tDCS is similarly effective than antidepressants would have a tremendous impact in clinical psychiatry, since tDCS is virtually absent of adverse effects. Its ease of use, portability and low price are also interesting characteristics for using in primary and secondary health care. Thus, our aim is to compare tDCS against a fully dosed, effective antidepressant. The study will be a non-inferiority, randomized, double-blinded, placebo-controlled, three-arm trial comparing active tDCS/placebo pill, sham tDCS/escitalopram 20mg/day and sham tDCS/placebo pill. Our primary aim is to show that tDCS is not inferior to escitalopram 20mg/day with a noninferiority margin of at least 50% of the escitalopram-placebo effect.

DETAILED DESCRIPTION:
Major depressive disorder (MDD) is a common psychiatric condition, mostly treated with antidepressant drugs, which are limited for issues such as refractoriness and adverse effects. In this context, the researchers investigate a non-pharmacological treatment known as transcranial direct current stimulation (tDCS). In a prior clinical trial with 120 patients with MDD, the investigators demonstrated that the combination of tDCS with sertraline 50mg/day had increased, faster effects on depressive symptoms (Brunoni et al., JAMA Psychiatry, 2013). However, although the investigators suggested that tDCS vs. sertraline had similar efficacy, such comparison was compromised due to the low sertraline dose and also because the comparison of sertraline vs. placebo was not significant. To prove that tDCS is similarly effective than antidepressants would have a tremendous impact in clinical psychiatry, since tDCS is virtually absent of adverse effects. Its ease of use, portability and low price are also interesting characteristics for using in primary and secondary health care. Thus, our aim is to compare tDCS against a fully dosed, effective antidepressant. The study will be a non-inferiority, randomized, double-blinded, placebo-controlled, three-arm trial comparing active tDCS/placebo pill, sham tDCS/escitalopram 20mg/day and sham tDCS/placebo pill for ten weeks, randomizing 240 patients with MDD in a 3:3:2 ratio (less to placebo). Our primary aim is to show that tDCS is not inferior to escitalopram 20mg/day with a noninferiority margin of at least 50% of the escitalopram-placebo effect. As secondary aims, the researchers will investigate putative biomarkers for tDCS response. This is important considering the large sample size of this study and also the paucity of tDCS studies - therefore, the identification of such biomarkers could generate new hypothesis for future studies and for tDCS' mechanisms of action. The biomarkers will be: genetic polymorphisms (BDNF, SLC6A4, THP1, 5HT2A); serum markers (BDNF); motor cortical excitability (cortical silent period, intracortical inhibition, intracortical facilitation); heart rate variability; and neuroimaging (structural volume of the dorsolateral prefrontal and anterior cingulate cortex, white matter tracts of the prefrontal cortex and posterior cingulate cortex connectivity). This project represents a novel research line in our Institution, and the investigators thereby propose the onset of a new center denominated C.I.N.A. (Interdisciplinary Center for Applied Neuromodulation) that will foment the use and development of projects using neuromodulation techniques. This new center will also interact with other centers on the fields of clinical research, neurosciences and neuropsychiatry.

ELIGIBILITY:
Inclusion Criteria:

* HAMD17>=17
* more than 8 years of schooling OR able to read, speak and understand the Portuguese language.
* Low suicide risk.

Exclusion Criteria:

* Bipolar disorders.
* Schizophrenia and other psychotic disorders.
* Anxiety disorders, if it is the primary diagnosis (comorbidity with depression is not an exclusion disorder)
* Substance abuse or dependence.
* Depression symptoms better explained by medical conditions.
* Neurologic conditions (e.g., stroke, multiple sclerosis, brain tumor).
* Severe medical conditions.
* Pregnancy/breast-feeding.
* Severe suicidal ideation, suicidal planning or recent (<4 weeks) suicide attempt.
* Contra-indications to escitalopram.
* Current use of escitalopram in the current depressive episode.
* Use of escitalopram in a prior depressive episode that was not effective.
* Contra-indications to tDCS.
* Previous use of tDCS (current or previous depressive episode).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2013-10; Primary Completion 2016-07 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Changes in Hamilton Rating Scale for Depression, 17 items (HAMD17) | Weeks 0 and 10
  Continuous measure (score changes). Non-inferiority assessment: the difference between tDCS to escitalopram should be >50% of escitalopram to placebo efficacy.

SECONDARY OUTCOMES:
Change in HDRS | Weeks 0, 3, 6, 8, 10
  Continuous measure (score changes).
Change in Montgomery-Asberg Depression Rating Scale (MADRS) | Weeks 0, 3, 6, 10
  Continuous measure (score changes).
Change in Beck Depression Inventory (BDI) | Weeks 0, 3, 6, 10
Change in Positive and Negative Affect Scale (PANAS) | Weeks 0, 3, 6, 10
Change in State-Trait Anxiety Inventory (STAI) | Weeks 0, 3, 6, 10
Hamilton Rating Scale for Depression, 17 items (HAMD17) | Week 10
  Response (≥50% improvement from week 0 to 10)
Hamilton Rating Scale for Depression, 17 items (HAMD17) | Week 10
  Remission (HAMD17 ≤7) at week 10.
Adverse events | Week 3 and Week 10.
  Assessment and comparisons of tDCS and drug adverse events. We used a tDCS adverse events questionnaire (Brunoni et al., 2011) and the SAFTEE.
Serious adverse events | Up to Week 10.
  Serious adverse events include treatment-emergent hypomania/mania (YMRS>8), suicide, psychiatric hospitalization and others life-threatening or incapacitant events.
Young Manic Rating Scale (YMRS) | Week 3 and Week 10.
  Assessment of treatment-emergent hypomania/mania, defined as YRMS>8.
Predictor of response | Week 10
  Age (years)
Predictor of response | Week 10
  Gender
Predictor of response | Week 10
  Low wage (less than 5 monthly wages in Brazil)
Predictor of response | Week 10
  Recurrent depression
Predictor of response | Week 10
  Chronic depression
Predictor of response | Week 10
  Refractory depression
Predictor of response | Week 10
  Severe depression
Predictor of response | Week 10
  Benzodiazepine use
Predictor of response | Week 10
  Higher education (>15 years of schooling)
Predictor of response | Week 10
  Age of onset of the depressive episode (years)
Predictor of response | Week 10
  Any anxiety disorder
Predictor of response | Week 10
  Physical activity
Predictor of response | Week 10
  melancholic depression
Predictor of response | Week 10
  atypical depression
Predictor of response | Week 10
  smoking status
Predictor of response | Week 10
  hypertension
Predictor of response | Week 10
  diabetes mellitus
Predictor of response | Week 10
  ethnicity
Predictor of response | Week 10
  marital status
Predictor of response | Week 10
  employment status
Predictor of response | Week 10
  obesity
Predictor of response | Week 10
  familial psychiatry history
Predictor of response | Week 10
  Temperament and Character Inventory - Novelty seeking
Predictor of response | Week 10
  Any tDCS related adverse event.
Predictor of response | Week 10
  Temperament and Character Inventory - Harm avoidance
Predictor of response | Week 10
  Temperament and Character Inventory - Reward Dependence
Predictor of response | Week 10
  Temperament and Character Inventory - Persistence
Predictor of response | Week 10
  Temperament and Character Inventory - Cooperativeness
Predictor of response | Week 10
  Temperament and Character Inventory - Self-transcendence
Predictor of response | Week 10
  Temperament and Character Inventory - Self-directedness
Predictor of response | Week 10
  FAS verbal fluency test
Predictor of response | Week 10
  Digit span forward
Predictor of response | Week 10
  Digit span backward
Predictor of response | Week 10
  Trail Making Test - A
Predictor of response | Week 10
  Trail Making Test - B
Predictor of response | Week 10
  Symbol digit
Predictor of response | Week 10
  Montreal Cognitive Assessment
Predictor of response | Week 3 and 10
  Motor Cortical Excitability - Cortical silent period (left and right hemispheres)
Predictor of response | Week 3 and 10
  Motor Cortical Excitability - Intracortical inhibition (left and right hemispheres)
Predictor of response | Week 3 and 10
  Motor Cortical Excitability - Intracortical facilitation (left and right hemispheres)
Predictor of response | Week 3 and 10
  Heart rate variability - HF
Predictor of response | Week 3 and 10
  Heart rate variability - LF
Predictor of response | Week 3 and 10
  Heart rate variability - RMSSD

CONTACTS AND LOCATIONS:
Overall Officials: Andre R Brunoni, MD, PhD, Principal Investigator — University of Sao Paulo
Locations (2):
- Brazil (2):
  - Hospital Universitário, Universidade de São Paulo, São Paulo, São Paulo
  - Institute of Psychiatry, HC-FMUSP, São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Goerigk SA, Padberg F, Chekroud A, Kambeitz J, Buhner M, Brunoni AR. Parsing the antidepressant effects of non-invasive brain stimulation and pharmacotherapy: A symptom clustering approach on ELECT-TDCS. Brain Stimul. 2021 Jul-Aug;14(4):906-912. doi: 10.1016/j.brs.2021.05.008. Epub 2021 May 26. PMID 34048940
- [Derived] Bulubas L, Padberg F, Bueno PV, Duran F, Busatto G, Amaro E Jr, Bensenor IM, Lotufo PA, Goerigk S, Gattaz W, Keeser D, Brunoni AR. Antidepressant effects of tDCS are associated with prefrontal gray matter volumes at baseline: Evidence from the ELECT-TDCS trial. Brain Stimul. 2019 Sep-Oct;12(5):1197-1204. doi: 10.1016/j.brs.2019.05.006. Epub 2019 May 8. PMID 31105027
- [Derived] Brunoni AR, Moffa AH, Sampaio-Junior B, Borrione L, Moreno ML, Fernandes RA, Veronezi BP, Nogueira BS, Aparicio LVM, Razza LB, Chamorro R, Tort LC, Fraguas R, Lotufo PA, Gattaz WF, Fregni F, Bensenor IM; ELECT-TDCS Investigators. Trial of Electrical Direct-Current Therapy versus Escitalopram for Depression. N Engl J Med. 2017 Jun 29;376(26):2523-2533. doi: 10.1056/NEJMoa1612999. PMID 28657871
- [Derived] Brunoni AR, Sampaio-Junior B, Moffa AH, Borrione L, Nogueira BS, Aparicio LV, Veronezi B, Moreno M, Fernandes RA, Tavares D, Bueno PV, Seibt O, Bikson M, Fraguas R, Bensenor IM. The Escitalopram versus Electric Current Therapy for Treating Depression Clinical Study (ELECT-TDCS): rationale and study design of a non-inferiority, triple-arm, placebo-controlled clinical trial. Sao Paulo Med J. 2015 May-Jun;133(3):252-63. doi: 10.1590/1516-3180.2014.00351712. Epub 2015 Jun 1. PMID 26176930
- See also: Trial information for participants and investigators. — http://www.sin.org.br